CLINICAL TRIAL: NCT04177680
Title: Pharmacodynamic Effects of a Free-fatty Acid Formulation of Omega-3 Pentaenoic Acid to ENHANCE Efficacy in Adults With Hypertriglyceridemia: The ENHANCE-IT Trial
Brief Title: Pharmacodynamic Effects of a Free-Fatty Acid Formulation of Omega-3 Pentaenoic Acid in Adults With Hypertriglyceridemia
Acronym: ENHANCE-IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Collaborators: Matinas Biopharma, Inc (Industry); MB Clinical Research and Consulting LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAT-002
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — MAT9001; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omega-3 pentaenoic acid (MAT9001) (Experimental): 2g MAT9001 capsules twice daily with meals
  Interventions: Drug: Omega 3 pentaenoic acid
- Icosapent ethyl (Vascepa) (Active Comparator): 2g Vascepa capsules twice daily with meals
  Interventions: Drug: icosapent ethyl

INTERVENTIONS:
Drug: Omega 3 pentaenoic acid — Encapsulated omega-3 pentaenoic acid
  Other Names: MAT9001
  Arms: Omega-3 pentaenoic acid (MAT9001)
Drug: icosapent ethyl — Encapsulated omega-3 acid ethyl esters
  Other Names: Vascepa
  Arms: Icosapent ethyl (Vascepa)

SUMMARY:
Pharmacodynamic effects of MAT9001 compared to Vascepa in adults with hypertriglyceridemia

DETAILED DESCRIPTION:
An open-label, randomized, crossover study to assess the pharmacodynamic effects of MAT-9001, an omega-3 free fatty acid compared to Vascepa (icosapent ethyl) on triglycerides and other lipoprotein lipids in men and women with elevated triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 y of age
* Judged to be in generally good health
* Fasting triglycerides ≥150 mg/dL to ≤499 mg/dL during screening
* Body mass index of ≥20.0 kg/m2
* No clinically significant findings in a 12-lead ECG or physical examination
* Willing and able to undergo the scheduled study procedures
* Understands study procedures and signs forms documenting informed consent to participate in the study

Exclusion Criteria:

* Laboratory test result of clinical significance
* Uncontrolled hypertension
* Clinically significant gastrointestinal, endocrine, cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic, or biliary disorder
* History of human immunodeficiency virus, hepatitis B or hepatitis C infection
* Used any medication intended to alter the lipid profile within 4 weeks of the first qualification visit
* Active systemic infection
* A condition the Investigator believes would interfere subject ability to provide informed consent and/or comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, Study Director — MB Clinical Research and Consulting
Locations (8):
- United States (8):
  - Matinas Investigational Site, Jacksonville, Florida
  - Matinas Investigational site, Jupiter, Florida
  - Matinas Investigational Site, Port Saint Lucie, Florida
  - Matinas Investigational Site, Addison, Illinois
  - Matinas Investigational Site, Chicago, Illinois
  - Matinas Investigational site, Indianapolis, Indiana
  - Matinas Investigational site, Louisville, Kentucky
  - Matinas Investigational site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maki KC, Bays HE, Ballantyne CM, Underberg JA, Kastelein JJP, Johnson JB, Ferguson JJ. A Head-to-Head Comparison of a Free Fatty Acid Formulation of Omega-3 Pentaenoic Acids Versus Icosapent Ethyl in Adults With Hypertriglyceridemia: The ENHANCE-IT Study. J Am Heart Assoc. 2022 Mar 15;11(6):e024176. doi: 10.1161/JAHA.121.024176. Epub 2022 Mar 1. PMID 35232215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study - each patient received both treatments
Groups:
- MAT9001 Then Vascepa: 2g MAT9001 capsules twice daily with meals for 4 weeks; 4 week washout; 2 g Vascepa (icosapent ethyl) twice daily with meals for 4 weeks
  Crossover design - Patients in this arm received initial treatment with MAT9001, a washout period, and treatment with Vascepa
- Vascepa Then MAT9001: 2g Vascepa (icosapent ethyl) twice daily with meals for 4 weeks; 4 week washout; MAT9001 2g twice daily with meals for 4 weeks
  Crossover design - Patients were randomized to receive initial treatment with Vascepa, a washout period, and treatment with MAT9001
Period: Overall Study
Arm/Group | MAT9001 Then Vascepa | Vascepa Then MAT9001
Started | 49 | 51
Completed | 47 | 48
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: All patients received both treatments
Arm/Group | Total Study Population
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 97
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] | 32.1 (6.6)
Lipid Drugs [Count of Participants; unit: Participants]
  Neither statin nor ezetimibe | 53
  Statin only | 46
  Both statin and ezetimibe | 1
Triglyceride stratification [Count of Participants; unit: Participants]
  < 2.26 mmol/L (< 200 mg/dL) | 41
  >= 2.26 - 5.64 mmol/l (200-499 mg/dL) | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Plasma Triglycerides (Pharmacodynamic Population)
Description: Percent change in triglycerides from baseline to end of treatment in the pharmacodynamic population
Time Frame: baseline to 28 days
Population: All patients with measurable results who received both drugs
Measure: Median (Inter-Quartile Range); unit: Percent Change from baseline
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
Number analyzed (Participants) | 94 | 94
Percent Change from baseline | -20.9 [-24.6 to -17.1] | -18.3 [-22.1 to -14.3]

2. Secondary Outcome: Percent Change in Other Plasma Lipoprotein Lipids (Pharmacodynamic Population)
Description: Percent change in other lipoprotein lipids from baseline to end of treatment in the pharmacodynamic population
Time Frame: baseline to 28 days
Population: All patients with measurable results who received both drugs
Measure: Median (Inter-Quartile Range); unit: Percent Change from baseline
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
Number analyzed (Participants) | 94 | 94
Percent Change from baseline
  Total Cholesterol | -5.6 [-7.3 to -3.8] | -4.1 [-5.9 to -2.3]
  Low density lipoprotein (LDL)-Cholesterol | -4.8 [-7.2 to -2.4] | -3.1 [-5.6 to -0.6]
  High density lipoprotein (HDL)-Cholesterol | -1.7 [-4 to 0.6] | -1.1 [-3.3 to 1.2]
  Very low density lipoprotein (VLDL)-Cholesterol | -15.5 [-18.3 to -12.5] | -13.3 [-16.2 to -10.3]
  non-HDL-Cholesterol | -7 [-9.1 to -4.8] | -5.2 [-7.4 to -3]

3. Secondary Outcome: Percent Change in Lipoprotein Lipids (Per Protocol Population)
Description: Percent change from baseline in lipoprotein lipids in the per protocol population
Time Frame: baseline to 28 days
Population: All patients who had measurable values for both treatments and had at least 80% compliance with study medication
Measure: Median (Inter-Quartile Range); unit: Percent Change from baseline
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
Number analyzed (Participants) | 82 | 82
Percent Change from baseline
  Triglycerides | -20 [-23.7 to -16.2] | -15.1 [-19 to -11]
  Total Cholesterol | -5.7 [-7.4 to -3.9] | -3.5 [-5.2 to -1.7]
  LDL-Cholesterol | -4.8 [-7.3 to -2.3] | -2.8 [-5.3 to -0.2]
  HDL-Cholesterol | -2.4 [-4.8 to 0] | -1.3 [-3.7 to 1.1]
  VLDL-Cholesterol | -15 [-17.8 to -12.1] | -10.9 [-13.8 to -7.8]
  Non-HDL-Cholesterol | -6.9 [-9 to -4.7] | -4.4 [-6.6 to -2.2]

4. Secondary Outcome: Percent Changes in Apolipoproteins, PCSK9 and Hs-CRP (Pharmacodynamic Population)
Description: The percent change from baseline in Apolipoproteins, PCSK9 and hs-CRP in the PD Population
Time Frame: baseline to 28 days
Population: All patients with measurable values who received both therapies
Measure: Median (Inter-Quartile Range); unit: Percent Change from baseline
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
Number analyzed (Participants) | 94 | 94
Percent Change from baseline
  Apolipoprotein (Apo) A1 | -4 [-5.6 to -2.3] | -3.1 [-4.7 to -1.5]
  Apo B | -3.5 [-5.9 to -1.1] | -2.5 [-4.9 to -0.2]
  Apo C3 | -12.4 [-15.8 to -9] | -11.1 [-14.4 to -7.7]
  Proprotein convertase subtilisin/kexin type 9 (PCSK9) | -6.6 [-10.9 to -2.1] | -7.3 [-11.5 to -2.9]
  High-sensitivity C-reactive protein (hs-CRP) | -5.8 [-15.3 to 4.7] | 8.5 [-2.4 to 20.7]

5. Secondary Outcome: Percent Change From Baseline in Omega-3 Fatty Acid Concentrations (Pharmacodynamic Population)
Description: The percent change from baseline in Omega-3 fatty acid concentrations in the Pharmacodynamic population
Time Frame: Baseline to 28 days
Population: Pharmacodynamic population - all patients with measurable values who received both drugs
Measure: Median (Inter-Quartile Range); unit: Percent Change from baseline
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
Number analyzed (Participants) | 94 | 94
Percent Change from baseline
  Eicosapentaenoic acid (EPA) | 848 [754 to 952] | 692 [614 to 778]
  Docosahexaenoic acid (DHA) | 1.7 [-2.0 to 5.5] | -3.3 [-6.8 to 0.2]
  Docosapentaenoic acid (DPA) | 177 [160 to 194] | 140 [126 to 155]
  EPA + DHA + DPA | 205 [187 to 225] | 165 [149 to 182]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over Treatment period 1 and Treatment period 2
Description: Adverse events were noted at each study visit while under treatment
Arm/Group | Omega-3 Pentaenoic Acid (MAT9001) | Icosapent Ethyl (Vascepa)
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/100
Other Adverse Events (participants affected / at risk) | 43/97 | 28/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 Pentaenoic Acid (MAT9001) (N=97) | Icosapent Ethyl (Vascepa) (N=100)
Total GI Disorders (Gastrointestinal disorders) | 25 | 11
Total Infections (Infections and infestations) | 4 | 2
Total Injury (Injury, poisoning and procedural complications) | 5 | 3
Total Musculoskeletal Disorders (Musculoskeletal and connective tissue disorders) | 7 | 7
Total Nervous System Disorders (Nervous system disorders) | 2 | 3
cataract (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 10 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Eructation (Gastrointestinal disorders) | 6 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 11 | 0
Urinary Tract infection (Infections and infestations) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04177680/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04177680/SAP_001.pdf